CLINICAL TRIAL: NCT01518322
Title: An Observational, Multi-Center, Single-Visit Study to Assess the Impact of FeNO Measured With the NIOX MINO® Device in Identifying Asthma Among Patients With Prolonged Respiratory Symptoms
Brief Title: Impact of FeNO Measured With the NIOX MINO® Device in Identifying Asthma Among Patients With Prolonged Respiratory Symptoms
Status: Completed | Type: Observational
Sponsor: Aerocrine AB (Industry)
Responsible Party: Sponsor
Other Study IDs: AER-040
Record Dates: First submitted 2011-11-11; First posted 2012-01-26 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-06

CONDITIONS: Asthma
Keywords: Asthma; Fractional Exhaled Nitric Oxide; Respiratory Symptoms; NIOX MINO; Inhaled corticosteroids; Nitric Oxide
MeSH Terms: conditions — Asthma; Signs and Symptoms, Respiratory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FeNO: All subjects will have their Fractional Exhaled Nitric Oxide (FeNO) measured with the NIOX MINO® device according to instructions for NO measurements.
  Interventions: Device: NIOX MINO®

INTERVENTIONS:
Device: NIOX MINO® — Fractional Exhaled Nitric Oxide (FeNO) will be measured with the NIOX MINO®

SUMMARY:
Overall Aim:

To better understand the diagnostic process for prolonged respiratory events and determine the potential role of FeNO in assessing the possibility of asthma as the symptoms etiology.

Study Objectives:

The specific objectives of this study are to:

* Determine the frequency of ICS prescription for the treatment of non-specific lower respiratory symptoms.
* Determine the frequency of asthma diagnosis as an etiology for the non-specific lower respiratory symptoms.
* Explore the value of FeNO in identifying asthma as the etiology of the non-specific lower respiratory symptoms.

Number of Subjects:

It is anticipated that up to approximately 3,000 patients will be asked to complete the brief screening questionnaire that will be used to identify up to approximately 280 eligible patients who meet the study inclusion/exclusion criteria during a (approximately) 4 to 6 week study enrollment period.

Reference Product: NIOX MINO®

Duration of the participants involvement in the investigation: Single Visit

Performance assessments:

Fractional Exhaled Nitric Oxide (FeNO) Measurements will be performed using the NIOX MINO® device according to "Instructions for NO measurements" which will be provided to each Investigative site prior to patient enrollment.

Safety Assessments:

The Investigator is responsible for the detection, reporting, and documentation of events meeting the definition of an Adverse Event (AE) and/or Serious Injuries as provided in this clinical investigation plan from the time of informed consent/assent and during the study period.

Criteria for Evaluation:

The relationship(s) between FeNO and both the diagnosis of asthma and prescription of ICS will be explored by correlation, measures of concordance and logistic modeling.

DETAILED DESCRIPTION:
INTRODUCTION:

Overview:

The measurement of exhaled nitric oxide (FeNO) is the only clinical test for measuring airway inflammation that can be performed consistently and accurately in clinical practice at the point-of-care. Airway inflammation is now recognized as the central mechanism in the pathogenesis of asthma and its symptoms. The measurement of FeNO with the NIOX MINO® device provides a rapid, noninvasive, and inexpensive tool to assess airway inflammation in asthma. The test is easy to perform and requires minimal training for the operator to conduct the test.

Burden of Disease:

The burden of asthma in the U.S. is significant and growing. In May 2011, the Centers for Disease Control and Prevention (CDC) reported that the prevalence of asthma has increased by 12.3% from 2001 to 2009 and affects approximately 24.6 million Americans, including 9.6% of the pediatric population. In 2008, at least one half (52.6%) of persons with asthma in the U.S. reported having an asthma attack in the preceding 12 months. In 2007, there were 1.75 million asthma-related emergency department visits and 456,000 asthma hospitalizations.

Initial assessment and diagnosis of asthma and ongoing management of asthma patients remain key challenges. The traditional approaches for diagnosing and management of asthma include family history evaluation, symptom assessment and airflow measures (e.g. spirometry). However, these approaches do not effectively incorporate measurement of inflammation into diagnosis and management approaches.

Role of Exhaled Nitric Oxide (FeNO):

FeNO has evolved as a predictive and prognostic biomarker for airway inflammation. Nitric oxide (NO) gas is produced in the epithelial cells of the bronchial wall as an intrinsic part of the inflammatory process.

Measuring the amount of FeNO is useful in the initial assessment of patients with chronic cough or symptoms suggestive of asthma, and for the management of patients on corticosteroid treatment. Exhaled nitric oxide increases when there is eosinophilic airway inflammation. Changes in FeNO precede changes in symptoms that are observed with increased and decreased airway inflammation. The measurement of FeNO is easily and rapidly accomplished, providing an objective, interpretable value that cannot be influenced by patient effort or variations in the clinician's test technique. FeNO measurement is a well-established and scientifically documented procedure with over 2000 publications on its use.

Intended Use:

NIOX MINO® measures Nitric Oxide (NO) in human breath. Nitric Oxide is frequently increased in some inflammatory processes such as asthma. The fractional NO concentration in expired breath (FeNO), can be measured by NIOX MINO with assurance that such measurements are repeatable and according to guidelines for NO measurement established by the American Thoracic Society.

Measurement of FeNO by NIOX MINO is a quantitative, non-invasive, simple and safe method to measure the decrease in FeNO concentration in asthma patients that often occurs after treatment with anti-inflammatory pharmacological therapy, as an indication of the therapeutic effect in patients with elevated FeNO levels. NIOX MINO is suitable for children, approximately 7 - 17 years, and adults 18 years and older.

Rationale for the Study:

The current study will generate information to characterize patients seeking health care in a Primary Care Clinic presenting with non-specific lower respiratory symptoms such as cough, wheeze, and/or shortness of breath that are associated with asthma but may be labeled as more acute respiratory conditions, e.g. infections. Results from this study may be used to estimate the number of patients required to demonstrate meaningful changes in non-specific lower respiratory symptoms in future studies and may also support the usefulness of FeNO in the Primary Care setting.

CLINICAL INVESTIGATION OBJECTIVES:

Overall Aim:

To better understand the diagnostic process for prolonged respiratory events and determine the potential role of FeNO in assessing the possibility of asthma as the symptoms etiology.

Study Objectives:

The specific objectives of this study are to:

* Determine the frequency of ICS prescription for the treatment of non-specific lower respiratory symptoms.
* Determine the frequency of asthma diagnosis as an etiology for the non-specific lower respiratory symptoms.
* Explore the value of FeNO in identifying asthma as the etiology of the non-specific lower respiratory symptoms.

CLINICAL INVESTIGATION PLAN:

Overall Clinical Investigation Design and Plan-Description:

An observational, multicenter, single-visit study to collect information on patients utilizing a Primary Care Clinic to seek health care for the assessment, treatment, and management of non-specific lower respiratory symptoms such as cough, wheeze, and/or shortness of breath. All patients seeking care at the clinic for any medical condition will be asked to complete a brief screening questionnaire designed to capture a self-assessment of non-specific lower respiratory symptoms. Patients with non-specific lower respiratory symptoms such as cough, wheeze, and/or shortness of breath who meet the inclusion/exclusion criteria for this study may be invited to participate in the study.

Visit and Procedures:

Subjects meeting Inclusion and Exclusion Criteria and who express interest in study participation will be asked to provide the following documentation and information: Informed Consent/Assent; Baseline Characteristics; Medical History

FeNO Measurement: A single blinded FeNO measurement will be obtained.

Patient Discharge from the Study: Once all information has been collected and procedures performed, the patient will be discharged from the clinic and their study participation will be complete.

Medical Record Review: Patient's medical record and administrative data will be reviewed before study close-out to assess the number of previous similar episodes each patient has had during the previous two (2) years.

Selection of Population:

Population Characteristics: Males and females, seven (7) to 65 years of age. It is anticipated that up to approximately 3,000 patients from multiple primary care clinics will complete the brief screening questionnaire that will be used to identify up to approximately 280 eligible patients who meet the study inclusion/exclusion criteria during a (approximately) 4 to 6 week study enrollment period.

Medical Device:

The NIOX MINO® was cleared by the FDA on March 4, 2008 as a new hand-held device for the measurement of exhaled Nitric Oxide, a marker of eosinophilic airway inflammation.

The NIOX MINO® is a 10 second test based on exhaled breath measured at a 50 ml/second flow rate. In this study the results will not be displayed, but will remain blinded to the investigator.

PERFORMANCE AND SAFETY ASSESSMENT:

Clinical performance assessments: Investigators should use their judgment to determine if study candidates will be able to successfully perform assessment of FeNO using the NIOX MINO®.

Clinical safety assessments: The Investigator is responsible for the detection, reporting, and documentation of events meeting the definition of an Adverse Event (AE) and/or Serious Injury as provided in this clinical investigation plan from the time of informed consent/assent and during the study period.

Adverse events:

* Adverse event: Any incident where the use of a medical device (including in vitro diagnostics) is suspected to have resulted in an adverse outcome in a patient.
* Serious injury: means injury or illness that:

  1. Is life-threatening, or
  2. Results in permanent impairment of a body function or permanent damage to a body structure, or
  3. Necessitates medical or surgical intervention to preclude permanent impairment of a body function or permanent damage to a body structure.
* Malfunction: the failure of a device to meet its performance specifications or otherwise perform as intended.
* Caused or contributed: the death or serious injury was or may have been attributed to a medical device, or that the medical device was or may have been a factor in a death or serious injury, including events occurring as a result of:

  1. Failure
  2. Malfunction
  3. Improper or inadequate design
  4. Manufacture
  5. Labeling
  6. User error

ELIGIBILITY:
Inclusion Criteria:

* Symptoms: Must have non-specific lower respiratory symptoms, such as cough, wheeze, and/or shortness of breath
* Age: Seven (7) to 65 years, inclusive
* Sex: Males and Females
* Ability to successfully perform assessment of FeNO: Investigators should use their judgment to determine if study candidates will be able to successfully perform assessment of FeNO using the NIOX MINO®.

Exclusion Criteria:

* Diagnosis: No previous or current diagnosis of asthma or chronic obstructive pulmonary disease (COPD).
* Medications: No use of inhaled or oral corticosteroids within 7 days prior to the visit.
* Study Participation Outside of This Protocol: Patients currently enrolled in studies of Investigational or non-Investigational Drugs or Medical Devices and/or who participated in these studies within 30 days prior to this study are excluded.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any person visiting a primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Herje, BSN, RN, MBA, Study Director — Aerocrine, Inc.; Barbara Yawn, MD, MSc, Principal Investigator — Olmsted Medical Center
Locations (13):
- United States (13):
  - Olmstead Medical Center Byron, Byron, Minnesota
  - Olmstead Medical Center Chatfield, Chatfield, Minnesota
  - Olmstead Medical Center Pine Island, Pine Island, Minnesota
  - Olmstead Medical Center Plainview, Plainview, Minnesota
  - Olmstead Medical Center Preston, Preston, Minnesota
  - Olmstead Medical Center Northwest, Rochester, Minnesota
  - Olmstead Medical Center - Allergy Department, Rochester, Minnesota
  - Olmstead Medical Center - Family Medicine Department, Rochester, Minnesota
  - Olmsted Medical Center - Internal Medicine Department, Rochester, Minnesota
  - Olmstead Medical Center St. Charles, Saint Charles, Minnesota
  - Olmstead Medical Center Spring Valley, Spring Valley, Minnesota
  - Olmstead Medical Center Stewartville, Stewartville, Minnesota
  - Olmstead Medical Center Wanamingo, Wanamingo, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 primary care clinics in the US. First Subject Enrolled: 01Nov2011. Last Subject Completed 16Feb2012.
Pre-assignment Details: Following completion of the screening questionnaire that collected information about self-reported non-specific lower respiratory complaints such as cough, wheeze or shortness of breath, eligible subjects were invited to participate in the study.
Period: Overall Study
Arm/Group | FeNO
Started | 235
Completed | 222
Not Completed | 13
Not completed — FeNO measurement was missing | 13

BASELINE CHARACTERISTICS:
Population: A total of 235 subjects were included in the All Subjects Population. 13 of the 235 subjects were missing the FeNO measurement.
Arm/Group | FeNO
Number analyzed (Participants) | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 211
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 40.9 (14.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 80
Region of Enrollment [Number; unit: participants]
  United States | 235

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between FeNO and the Diagnosis of Asthma
Description: For the primary analysis, the total number of subjects diagnosed with asthma is tabulated by Fractional Exhaled Nitric Oxide (FeNO). FeNO is split into high, intermediate and low categories and the associated kappa statistics and 95% confidence intervals are presented. FeNO grouping will be calculated per the American Thoracic Society (ATS) standards. For children under age 12 years, <20 ppb is low, ≥20 ppb and ≤35 ppb is intermediate, and >35 ppb is high. For those aged 12 years or older, <25 ppb is low, ≥25 ppb and ≤50 ppb is intermediate, and >50 ppb is high.
Time Frame: Single-visit, one (1) FeNO measurement. One (1) timepoint (Day 1)
Population: A total of 235 subjects were initially deemed eligible for the study and were identified as the All Subjects Population. Following review of the eligibility criteria and FeNO, 73 subjects were excluded from the Per Protocol Population, predominantly because of their prior asthma and COPD history and missing FeNO values.
Measure: Number; unit: participants
Groups:
- Low FeNO: Subjects with their Fractional Exhaled Nitric Oxide (FeNO) measured with the NIOX MINO® device according to instructions for NO measurements and Low FeNO per the American Thoracic Society (ATS) standards. For children under age 12 years, <20 ppb is low. For those aged 12 years or older, <25 ppb is low.
- Intermediate FeNO: Subjects with their Fractional Exhaled Nitric Oxide (FeNO) measured with the NIOX MINO® device according to instructions for NO measurements and intermediate FeNO per the American Thoracic Society (ATS) standards. For children under age 12 years, ≥20 ppb and ≤35 ppb is intermediate. For those aged 12 years or older, ≥25 ppb and ≤50 ppb.
- High FeNO: Subjects with their Fractional Exhaled Nitric Oxide (FeNO) measured with the NIOX MINO® device according to instructions for NO measurements and High FeNO per the American Thoracic Society (ATS) standards. For those aged 12 years or older, >50 ppb is high. For children under age 12 years, >35 ppb is high.
Arm/Group | Low FeNO | Intermediate FeNO | High FeNO
Number analyzed (Participants) | 98 | 42 | 22
participants | 1 | 1 | 1
Statistical Analysis 1: Comparison: Low FeNO vs Intermediate FeNO vs High FeNO; Kappa statistics were used to determine the level of agreement between FeNO measurements and asthma diagnosis using the a dichotomous schemes a measurement greater than 35 ppb for children under the age of 12 years or greater than 50 ppb for subjects at least 12 years of age was considered high; Test type: Superiority or Other; Kappa Statistics = 0.0490, 95% CI 2-sided [-0.0895 to 0.1875]

2. Primary Outcome: Relationship Between FeNO and the Prescription of ICS in Primary Care Practices
Description: The total number of subjects prescribed Inhaled Corticosteroids (ICS) will be tabulated by Fractional Exhaled Nitric Oxide (FeNO). FeNO is split into high, intermediate and low categories and the associated kappa statistics and 95% confidence intervals are presented. FeNO grouping will be calculated per the American Thoracic Society (ATS) standards. For children under age 12 years, <20 ppb is low, ≥20 ppb and ≤35 ppb is intermediate, and >35 ppb is high. For those aged 12 years or older, <25 ppb is low, ≥25 ppb and ≤50 ppb is intermediate, and >50 ppb is high.
Time Frame: Single-visit, one (1) FeNO measurement. One (1) timepoint (Day 1)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Low FeNO | Intermediate FeNO | High FeNO
Number analyzed (Participants) | 98 | 42 | 22
participants | 5 | 1 | 0

3. Secondary Outcome: Subjects With a History of Cough, Wheeze, and/or Shortness of Breath Prior to the Study
Description: The total number of subjects who reported prior episodes of cough, wheeze, and shortness of breath.
Time Frame: anytime prior to the single study visit
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Low FeNO | Intermediate FeNO | High FeNO
Number analyzed (Participants) | 98 | 42 | 22
participants | 65 | 25 | 13

4. Post Hoc Outcome: Of the 22 Subjects With a High FeNO (>50ppb Age 12 Years and Above; >35ppb Age Less Than 12 Years)During the Original Study Visit, Number of Subjects Subsequently Treated With Asthma Medications or Diagnosed With Asthma.
Description: A medical record review of the 22 subjects with a high FeNO Value (>50ppb age 12 years and above; >35ppb age less than 12 years)during the original study visit was conducted. The number of subjects who were either diagnosed with asthma or treated with asthma medications is presented.
Time Frame: 4 to 6 months after the original study visit.
Population: Of the 162 subjects in the per-protocol population, 22 had a high FeNO (>50ppb age 12 years and above; >35ppb age less than 12 years). A retrospective medical record review was conducted and the number of subjects either diagnosed with asthma or treated with asthma medications is presented.
Measure: Number; unit: participants
Arm/Group | High FeNO
Number analyzed (Participants) | 22
participants | 5

ADVERSE EVENTS:
Arm/Group | FeNO
Serious Adverse Events (participants affected / at risk) | 0/235
Other Adverse Events (participants affected / at risk) | 0/235

LIMITATIONS AND CAVEATS:
Physicians were blinded to FeNO results during the study, therefore asthma diagnoses and ICS prescriptions were made without knowledge of FeNO results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less